CLINICAL TRIAL: NCT01615432
Title: Comparison of Four Different Ventilators for Noninvasive Ventilation in Terms of Patient-ventilator Synchrony and Comfort
Brief Title: Comparison of Synchrony Between 4 NIV Ventilators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Prof. Philippe Jolliet, Main investigator, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Synchro_Non invasive vent
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Respiratoy Failure Requiring NIV Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: V-PAP III ventilator
Device: Stellar 150 ventilator
Device: BiPAP vision ventilator
Device: V60 ventilator

SUMMARY:
Comparison of the effects of 4 ventilators dedicated to NIV (2 home ventilators and 2 ventilators designed for NIV) on patient-ventilator synchrony and comfort in patients admitted in the intensive care unit for respiratory failure and treated with NIV.

ELIGIBILITY:
Inclusion Criteria:

* respiratory failure

Exclusion Criteria:

* Severe hypoxemia requiring an FiO2 > 0.6
* Hemodynamic instability : defined as a variation of > 20% in mean arterial pressure (MAP) and heart rate (HR) during the previous 2 hours; the need for high doses of catecholamines (namely > 0.5 mcg/kg/min) and/or the need of major volume resuscitation (more than 2 liters of fluids in 2 hours)
* Impaired consciousness or absence of patient cooperation;
* Facial or laryngeal lesions contraindicating the use of NIV;
* Poor short term prognosis.
* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Patient-ventilator synchrony
  Patient-ventilator synchrony will be assessed breath by brath on the basis of airway pressure, flow and diaphragmatic electrical activity recordings.

SECONDARY OUTCOMES:
comfort of patient under NIV
  Patient's confort during NIV will be assessed using a visual analogic scale.
Ventilatory parameters
  Tidal volume, respiratory rate, inspiratory time, expiratory time and maximal and mean airway pressure will be measured from the continuous recording of airway pressure and flow.

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive care and burn unit / CHUV, Lausanne, Canton of Vaud, Switzerland